CLINICAL TRIAL: NCT02772328
Title: Randomized Controlled Trial of a Social-network Oriented Mobile Health Based Intervention to Increase Access and Adherence to Hepatitis C Treatment and HIV Viral Suppression
Brief Title: A Peer-based Mobile-health Intervention to Increase Access & Adherence to Hepatitis C Treatment & HIV Viral Suppression
Acronym: HCV-TTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 1R01DA040488 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Hepatitis C; HIV; Risk Reduction Behavior
Keywords: Testing; Access
MeSH Terms: conditions — Hepatitis C; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peer Mentor (Experimental): Individuals in this arm will be trained in communication skills to promote HIV and HCV testing to their social network members, linkage to care and risk reduction behaviors.
  Interventions: Behavioral: Peer Mentor
- Neighborhood Matters (No Intervention): Participants in this arm will view a 15-20 minute video on issues in neighborhoods such as crime and violence, restoring communities and incarceration and discuss their reactions and thoughts.

INTERVENTIONS:
Behavioral: Peer Mentor — comparison of communication training to equal attention control
  Arms: Peer Mentor

SUMMARY:
The purpose of this study is to test an intervention designed to train persons who inject drugs (PWID) and are infected with hepatitis C (HCV) and HIV in communication skills to 1) promote new HCV treatment and care 2) risk reduction and 3) recruit their social network members for HIV and HCV testing and linkage to care.

DETAILED DESCRIPTION:
The investigators propose recruiting 300 HIV/HCV co-infected PWID (i.e. Index participants). Half will be randomly assigned to the experimental condition and half to the equal attention comparison. The experimental intervention will include 8 group sessions that focus on communication to social network members, medical adherence and risk reduction skills, 2 dyad sessions with network members, monthly booster sessions for 6 months, and mHealth cuing of behavior for 6 months. These Index participants will be followed for 24 months (3, 6, 12, 18, & 24 month assessments). Participants who test positive for HCV will be linked to the Johns Hopkins Viral Hepatitis clinic to assess liver function and HCV chronicity and if applicable offered HCV treatment. Additionally, 450 network members will be recruited and will be tested for HIV and HCV and followed longitudinally to examine the social diffusion and social network factors associated with adherence among the Index participants.

ELIGIBILITY:
Inclusion Criteria:

* HCV antibody positive
* HIV antibody positive
* lifetime history of injection drug use
* interrupted HIV care:>3 months since HIV care or detectable viral load
* willingness to participate in group sessions and have conversations with social network members

Exclusion Criteria:

- participated in a behavioral intervention in prior 2 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Continuity in HIV care scale | 24 months
Access to HCV care scale | 24 months
  Initiation of HCV care at a viral hepatitis clinic

SECONDARY OUTCOMES:
HIV medication adherence scale | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Carl A Latkin, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Karin E Tobin, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Lighhouse Studies @ Peer Point, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will work with NIH to determine sharing plan